CLINICAL TRIAL: NCT04175015
Title: The SMARTY Trial: Evaluating the Effects of Colour of Candy on Perceptions of Taste. A Randomised Trial
Brief Title: The SMARTY Trial: Evaluating the Effects of Colour of Candy on Perceptions of Taste
Acronym: SMARTY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not feasible to randomise participants due to the logistics of the science festival at which we were planning to run the trial.
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Prof. Declan Devane, Scientific Director, HRB-Trials Methodology Research Network, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NUIreland-SMARTY
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Education
Keywords: Education; Randomised trial; Children; SMARTY
MeSH Terms: interventions — Candy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single - Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants will be randomised to eat an orange coloured smartie©
  Interventions: Other: Smartie© sweet/candy
- Control Group (Active Comparator): Participants will be randomised to eat a pink coloured smartie ©
  Interventions: Other: Smartie© sweet/candy

INTERVENTIONS:
Other: Smartie© sweet/candy — one chocolate sweet/ chocolate candy

SUMMARY:
The purpose of this trial is to determine if the colour of sweets (candy) effects taste.

DETAILED DESCRIPTION:
The purpose of this trial is to increase children's awareness of randomised controlled trials and gain insights into the best way to conduct a fair comparison. Everyday children are faced with health claims, some reliable and some not so reliable. The purpose of the SMARTY trial is to help children critically assess and develop a critical eye when it comes to information they encounter every day, in particular when it comes to their health. The SMARTY trial is a pragmatic, two group, parallel, randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* parental/guardian consent obtained

Exclusion Criteria:

* unable or unwilling to ingest intervention.
* medical conditions which prohibit ingestion of intervention (ie allergy, intolerance etc)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-24 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
Taste | 15 minutes
  Participants will be asked to indicate on visual scale how much they like the taste of the smartie© they ate using the 'single-item sleep quality scale (SQS)' . The SQS is a self-administered visual analogue scale on which respondents rate the overall quality of sleep over a 7-day recall period on a likert type scaling option from 0 to 10, according to the following five categories: 0 = terrible, 1-3 = poor, 4-6 = fair, 7-9 = good, and 10 = excellent .

CONTACTS AND LOCATIONS:
Overall Officials: Declan Devane, PhD, Principal Investigator — National University of Ireland, Galway
Locations (1):
- National University of Ireland Galway, Galway, Co. Galway, Ireland

IPD SHARING:
Plan to Share IPD: No